CLINICAL TRIAL: NCT05896956
Title: The Construction of Clinical Database and Multiomics Biobank Based on a Multicentral Prospective Cohort of Benign and Malignant Biliary Tract Diseases 胆道系统良恶性肿瘤前瞻性登记队列数据库与多组学生物样本库建设
Brief Title: The Construction of Clinical Database and Multiomics Biobank Based on a Multicentral Prospective Cohort of Benign and Malignant Biliary Tract Diseases
Status: Not yet recruiting | Type: Observational
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, Liu Ying-bin, Prof., RenJi Hospital
Other Study IDs: CRGGCpros
Record Dates: First submitted 2023-06-01; First posted 2023-06-09 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-06

CONDITIONS: Biliary Tract Diseases; Gallbladder Cancer; Extrahepatic Bile Duct Cancer; Intrahepatic Cholangiocarcinoma; Biliary Tract Neoplasms; Gall Stone
Keywords: biliary tract diseases; gallbladder cancer; biliary tract neoplasms; biliary tract cancer; cohort study
MeSH Terms: conditions — Biliary Tract Diseases; Gallbladder Neoplasms; Bile Duct Neoplasms; Cholangiocarcinoma; Biliary Tract Neoplasms; Gallstones

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with benign or malignant tumors of the biliary system: Patients enrolled should be clinically diagnosed with benign or malignant tumors of the biliary system, including unoperated patients with preliminary diagnosis of benign or malignant tumors of the biliary tract based on imaging examinations and laboratory test results, or pathological examination of patients treated with surgery confirmed as benign and malignant tumors of the gallbladder; The primary tumor is located in the extrahepatic bile ducts, intrahepatic bile ducts, gallbladder floor, gallbladder body, gallbladder neck, or gallbladder duct.
  Interventions: Other: no interventions

INTERVENTIONS:
Other: no interventions — no interventions

SUMMARY:
The aim of the study is to establishing a standardized biobank and a clinical information database for patients with benign and malignant tumors of the biliary system. With follow-up plans and advanced multiomics technology, a multiomics database for patients with benign and malignant tumors of the biliary tract will be further established. Based on the above work, real-world clinical research on the diagnosis and treatment of biliary tract tumors is about to be carried out, and a high-standard cohort research foundation is laid for precision therapy based on multiomics characteristics and molecular typing of biliary tract tumors.

DETAILED DESCRIPTION:
1. Trial population From the date of commencement of the study, patients who presented to the participating medical institutions in the study and were clinically diagnosed as benign or malignant tumors of the biliary system, and who met the inclusion criteria and did not meet any of the exclusion criteria, were enrolled in the study cohort after signing an informed consent form.

Diagnostic criteria:

Patients with benign biliary tumors and biliary malignant tumors diagnosed by pathology, and combined with clinical manifestations and imaging results, the first diagnosis and discharge were diagnosed as patients with advanced biliary malignant tumors.

Inclusion Criteria:

1. Sign informed consent, have good compliance, and be willing to accept follow-up and provide blood samples
2. Age 18-74 years old, gender is not limited
3. Clinical diagnosis of benign and malignant tumors of the biliary system, including unoperated patients preliminarily diagnosed as benign and malignant tumors of the biliary tract according to the results of imaging examinations and laboratory tests, or pathological examination of patients treated with surgery confirmed as benign and malignant tumors of the gallbladder
4. The primary tumor is located in the extrahepatic bile duct, intrahepatic bile duct, gallbladder floor, gallbladder body, gallbladder neck or gallbladder duct
5. Karnofsky performance score greater than 50

Exclusion Criteria:

1. Patients with biliary malignant tumors, biliary malignant tumor foci are not primary lesions.
2. Patients with biliary malignant tumors, combined with serious central nervous system diseases, respiratory diseases, autoimmune diseases, chronic renal insufficiency and other diseases, long-term use of immunosuppressants, combined with serious uncontrolled infections
3. Patients with biliary malignant tumors, who also have active cardiovascular and cerebrovascular diseases, have cerebrovascular accidents, myocardial infarction, unstable angina pectoris, or grade II. or above congestive heart failure according to the standards of the New York Heart Association, and require serious arrhythmias requiring drug treatment
4. Patients with biliary malignant tumors, women of childbearing age who have a positive blood pregnancy test or have not had a pregnancy test, pregnant or breastfeeding women
5. The patient is participating in other therapeutic clinical trials where treatment measures cannot be clarified or treatment information cannot be collected 2. Sample size calculation In this study, based on the retrospective cohort statistics of CRGGC study, the average number of gallbladder cancer patients admitted to the hospital in previous years, and the proportion of gallbladder cancer to biliary malignant tumors in previous epidemiological investigations, the number of potential research subjects actually diagnosed and treated by each participating unit was estimated, and the study sample size was calculated. The number of cases of benign and malignant biliary tumors included in the cohort of benign and malignant tumors of the biliary tract in this study is expected to reach 60% of the total number of hospitalized patients admitted by the participating units every year, and it is expected that no less than 250 patients with benign and malignant tumors of the biliary tract will be enrolled every year, and 500 patients are expected to be enrolled within a baseline period of 2 years from the date of the start of the study.

3. Specific research content The target population of this study is patients with benign and malignant tumors of the biliary system, and the potential sample group is patients diagnosed with benign and malignant tumors of the biliary system in the participating medical institutions since December 31, 2022 and meet the criteria for inclusion and exclusion of the study, and based on the retrospective cohort statistics of the CRGGC study, the average number of patients with gallbladder cancer admitted to the hospital in previous years, as well as the proportion of gallbladder cancer to biliary malignant tumors in previous epidemiological investigations, the number of potential research subjects actually diagnosed and treated by each participating unit was estimated. Calculate the study sample size. The number of cases of benign and malignant biliary tumors included in the cohort of benign and malignant tumors of the biliary tract in this study is expected to reach 60% of the total number of hospitalized patients admitted by the participating units every year, and it is expected that no less than 250 patients with benign and malignant tumors of the biliary tract will be enrolled every year, and 500 patients are expected to be enrolled within a baseline period of 2 years from the date of the start of the study. This study cohort is a single-disease registry cohort, which does not involve grouping at the stage of establishing the registration cohort, but in the data analysis stage, it can be divided into different subgroups such as biliary malignant tumors, benign biliary tumors, gallbladder cancer, intrahepatic cholangiocarcinoma, and extrahepatic cholangiocarcinoma according to the diagnosis of the included patients.

The research objectives of this study mainly include: (1) establishing a structured special disease dataset standard for biliary tumors based on the diagnosis and treatment norms and clinical pathways of biliary tract tumors; (2) Carry out clinical registration research on biliary tumors and build a special disease cohort; (3) Establish a biobank of biliary tumor cohort, including clinical diagnosis and treatment information such as patient diagnosis, surgery, treatment, progression, survival, and biological samples such as tumor tissue and body fluids; (4) Formulate standard operating specifications and sample quality control plans for the collection, transportation, acceptance, preparation, preservation and detection of biliary tumor biological specimen banks; (5) Formulate unified specimen bank management standards and information and data management processes, promote the intelligent management of specimen banks, and realize the linkage and integration of biobanks and specialized disease cohort databases; (6) Combine biliary tumor database, biomics technology, such as genomics, transcriptomics, proteomics, metabolomics technology, and big data acquisition, storage analysis technology to complete the molecular typing of biliary tumors.

The outcome indicators of this study included overall survival time OS, recurrence-free survival time PFS, R0 resection rate of patients treated with biliary malignancy, and objective response rate ORR. The main measurement indicators of this study include the patient's demographic information, past history, life history, admission, preoperative examination information, surgery, postoperative situation, discharge, follow-up, outcome indicators, routine examination results of biological samples and multi-omics sequencing results, the above data are derived from the original records of prospective case questionnaires, the original records of patients' electronic medical records and the examination results of patients' biological samples. The outcome of follow-up was defined as patients having been followed up for five years, or having a patient lost to follow-up or dying during follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Sign informed consent, have good compliance, and be willing to accept follow-up and provide blood samples.
2. Age 18-74 years old, gender is not limited.
3. Clinical diagnosis of benign and malignant tumors of the biliary system, including unoperated patients preliminarily diagnosed as benign and malignant tumors of the biliary tract according to the results of imaging examinations and laboratory tests, or pathological examination of patients treated with surgery confirmed as benign and malignant tumors of the gallbladder.
4. The primary tumor is located in the extrahepatic bile duct, intrahepatic bile duct, gallbladder floor, gallbladder body, gallbladder neck or gallbladder duct.
5. Karnofsky performance score greater than 50.

Exclusion Criteria:

1. Patients with biliary malignant tumors, biliary malignant tumor foci are not primary lesions.
2. Patients with biliary malignant tumors, combined with serious central nervous system diseases, respiratory diseases, autoimmune diseases, chronic renal insufficiency and other diseases, long-term use of immunosuppressants, combined with serious uncontrolled infections.
3. Patients with biliary malignant tumors, who also have active cardiovascular and cerebrovascular diseases, have cerebrovascular accidents, myocardial infarction, unstable angina pectoris, or grade II. or above congestive heart failure according to the standards of the New York Heart Association, and require serious arrhythmias requiring drug treatment.
4. Patients with biliary malignant tumors, women of childbearing age who have a positive blood pregnancy test or have not had a pregnancy test, pregnant or breastfeeding women.
5. The patient is participating in other therapeutic clinical trials where treatment measures cannot be clarified or treatment information cannot be collected.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with benign biliary tumors and biliary malignant tumors diagnosed by pathology, and combined with clinical manifestations and imaging results, the first diagnosis and discharge were diagnosed as patients with advanced biliary malignant tumors.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
overall survival | The last follow-up ended with the first of all patients followed up to death, loss to follow-up or withdrawal of informed consent, or follow-up for 2 years.
  OS in patients with biliary malignancies was long-term follow-up data, defined as the primary endpoint, OS is calculated from the date of surgery for patients treated surgically, and OS is calculated from the date of diagnosis for patients treated non-surgically. The expected survival of patients with benign biliary tumors is longer, and this study does not select the study endpoint based on the follow-up of patients with benign biliary tumors, but mainly collects perioperative diagnosis and treatment data and collects biological samples.

SECONDARY OUTCOMES:
progression-free survival | The last follow-up ended with the first of all patients followed up to death, loss to follow-up or withdrawal of informed consent, or follow-up for 2 years.
  PFS was defined as a secondary endpoint. PFS is calculated from the date of surgery for patients treated surgically, and PFS is calculated from the date of diagnosis for patients treated non-surgically. The expected survival of patients with benign biliary tumors is longer, and this study does not select the study endpoint based on the follow-up of patients with benign biliary tumors, but mainly collects perioperative diagnosis and treatment data and collects biological samples.

CONTACTS AND LOCATIONS:
Overall Officials: Ying-Bin Liu, PhD, Principal Investigator — RenJi Hospital